CLINICAL TRIAL: NCT05483569
Title: The Effect of Multidimensional Diaphragmatic Breathing Exercises and Fascial Release Techniques on the Treatment of Lower Extremity Lymphedema Caused by Gynecological Cancer Treatment
Brief Title: Diaphragmatic Exercises and Fascial Release Techniques on the Treatment of Lower Extremity Lymphedema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Ayca Evkaya Acar, Lecturer, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/0406
Record Dates: First submitted 2022-07-29; First posted 2022-08-02 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Lower Extremity Lymphedema
Keywords: Lower Extremity Lymphedema; Diaphragmatic Breathing Exercises; Fascial Release Techniques; Gynecological Cancer Treatment

STUDY DESIGN:
Intervention Model Description: There will be two groups in this study. Each group will consist of 15 women aged 25-65 years with Lower Extremity Lymphedema Caused by Gynecological Cancer Treatment. A total of 30 participants will take part in the study. CDP program and placebo fascial release techniques will be applied to the participants in Group 1 and, in addition to the CDP program, the participants in Group 2 will be given multidimensional diaphragmatic breathing exercises and fascial release techniques will be applied.
Who Masked: Outcomes Assessor
Masking Description: Participants will be divided into two groups using the block randomization method. Participants will be randomly distributed into 2 blocks of 15 participants. Each group using random number generation technique by computer. All evaluations will be made by the researcher who did not participate in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complex Decongestive Physiotherapy (Other): CDP program consisting of 4 parameters will be applied to this group. These parameters are MLD, Skin care, Multi-layer bandage application and decongestive exercises. In addition, the Placebo Facial Release technique will be performed by keeping the physiotherapist's hand in contact with the patient's abdominal region without applying any pressure and tension during the breathing exercises. Participants will be treated for a total of 3 weeks, 5 days a week. Each treatment session will last 45 minutes.
  Interventions: Other: Complex Decongestive Physiotherapy
- Multidimensional Diaphragmatic Breathing Exercises and Facial Release Technique (Experimental): CDP program consisting of 4 parameters will be applied to this group. These parameters are MLD, Skin care, Multi-layer bandage application and decongestive exercises. In addition, Multidimensional Diaphragmatic Breathing Exercises and Facial Release technique will be applied. These two treatments consist of these sub-exercises. These; Mechanical nose opening techniques, Intermittent Sniffing exercise, Diaphragm Awareness and Exercise Short Protocol, Thorax mobilization exercises, Myofascial diaphragm release techniques, Myofascial release exercises and postures and, Pelvic floor myofascial release postures.
  Participants will be treated for a total of 3 weeks, 5 days a week. Each treatment session will last 45 minutes.
  Interventions: Other: Multidimensional Diaphragmatic Breathing Exercises; Other: Facial Release Technique

INTERVENTIONS:
Other: Complex Decongestive Physiotherapy — Complete or complex decongestive physiotherapy (CDP) is a treatment for lymphedema, a condition in which excess fluid (lymph) collects in a part of the body. Damage to the lymph nodes or vessels, or a blockage leading to chronic swelling, usually causes lymphedema.
  Arms: Complex Decongestive Physiotherapy
Other: Multidimensional Diaphragmatic Breathing Exercises — Diaphragmatic breathing is an exercising technique to help strengthen your diaphragm and fill your lungs with air more efficiently.
  Arms: Multidimensional Diaphragmatic Breathing Exercises and Facial Release Technique
Other: Facial Release Technique — Fascial release is a manual therapy method that is applied holistically to the muscles and surrounding fascia through mechanical stimulation. It is a comprehensive approach to the evaluation and treatment of the muscular and fascia system in the body.
  Arms: Multidimensional Diaphragmatic Breathing Exercises and Facial Release Technique

SUMMARY:
The aim of this study is to determine the effect of multidimensional breathing exercises and fascial release techniques performed in addition to the conventional treatment program on the treatment of lymphatic fluid in women with lower extremity lymphedema due to gynecological cancer treatment, and the reflection of these practices on the functional level, sleep and quality of life.

DETAILED DESCRIPTION:
Secondary lower extremity lymphedema is frequently encountered after gynecological (endometrial, cervical, ovarian, vulvar/vaginal) cancer treatments. Lymphedema is a non-curative disease that is characterized by fluid and protein accumulation in the subcutaneous space. In the later stages, secondary skin changes and ulcers accompany, but it can cause complications such as fatigue, decrease in physical activity level, sleep and sexual dysfunction, and decrease in quality of life. Depending on the damaged area of the lymphatic system, it is exposed unilaterally or bilaterally, and in some cases, it also covers the lower body quarter and genital area. Chemotherapy and radiotherapy applications are a factor in its emergence. However, it has been reported that the main cause of lymphedema associated with gynecological cancer is the intervention in abdominal lymph nodes (para-aortic/-caval/external iliac/obturator/internal iliac/common iliac/presacral) and inguinal lymph nodes, especially pelvic. Studies have shown that lymph node interventions disrupt lymphatic flow and the risk of lymphedema exposure increases in direct proportion to the number of lymph nodes removed.

The superficial lymphatic drainage of the lower extremity occurs through lymphatic collectors, mainly to the inguinal and to a lesser extent, to the popliteal region lymph nodes. Lymph fluid passing through the deep lymphatic system from these regions, follows the pelvic lymph nodes, lumbar lymph nodes, lumbar trunks, cisterna chyli, and ductus thoracicus, respectively, and discharges into the venous system from the left venous aspect. Because of its passage through the abdominal and thoracic cavities, lower extremity lymphatic drainage is affected by thoracolumbal diaphragmatic motility. It has been reported that diaphragmatic movement creates positive pressure in the abdominal region during inspiration, providing the filling of lymph collectors/nodules (also venous system) in this region. On the other hand, negative pressure in the thoracic region during expiration results in a vacuum effect that accelerates the flow in the lend nodule and collectors towards the venous angle in both the thoracic and abdominal regions. The fact that approximately 60% of the lymph nodes in the body are below the diaphragm and the presence of a unique lymphatic drainage area on the peritoneal surface of the diaphragm shows how high the contribution of diaphragmatic movement to lymphatic drainage is.

Effectively fulfilling the function of the diaphragm (respiratory and veno-lymphatic drainage); It has been reported that it depends on the position and range of motion of the diaphragm. The position of the diaphragm is defined by the Zone of Apposition (ZOA) (the distance between the insertion of the diaphragm and its apex).

The shorter/longer than normal length of this area, which normally represents 30% of the total costal surface, is defined as the "suboptimal position". Suboptimal position indicates that the movement of the diaphragm is not optimal. Among the factors that cause suboptimal position of ZOA, somatic disorders and impaired posture are shown in the first place. In addition, it has been reported that the diaphragm is associated with many structures in the abdominal region via the fascia, and the fascial mobility of the abdominal region affects the position and movement of the diaphragm. In addition, it has been reported that the pelvic floor (pelvic diaphragm) opens in parallel with the movement of the thoracolumbal diaphragm, playing a role in controlling the intra-abdominal pressure during inspiration and contributing to the expansion of the limits of the mobility of the diaphragm. All these factors suggest that they may be associated with normalizing the mobility of the abdominal fascia and pelvic diaphragm in order to optimize the position and mobility of the diaphragm, thereby maximizing its function.

Lymphedema treatment is generally performed with Complex Decongestive Physiotherapy (CDP), which is offered as the most valid method by the International Society of Lymphology (ISL) and consists of manual lymph drainage (MLD), skin care, multi-layer bandage application and exercise. In manual lymph drainage, the fluid in the lymphedema area is sent to the nearest healthy absorption areas by using anastomosis routes. Although breathing exercises are performed in the exercise section of the CDP, multidimensional breathing exercises and fascia release applications to optimize the movement of the diaphragm (increasing the movement of the diaphragm, abdominal fascia and pelvic diaphragm) are not used. Investigators think that increasing the working performance of healthy collectors and nodules with applications that optimize the position and mobility of the diaphragm (which may be impaired due to surgical interventions and/or radiotherapy applications) will support impaired thoraco-abdominal lymphatic flow due to interventions for gynecological cancer (radiotherapy and lymph node dissection). The aim of this study is to investigate the effect of multidimensional diaphragmatic breathing exercises and abdominal fascial release techniques on the treatment of lower extremity lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 25-65
* Having unilateral lower extremity lymphedema (including/not including the trunk) due to gynecological cancer diagnosis and treatment method.
* Having Stage 1 and 2 lymphedema according to the International Society of Lymphology (ISL) classification
* Having situation that prevents the application of manual lymph drainage (cardiac edema, acute deep vein thrombus, acute renal failure, acute pulmonary edema, etc.)
* Having a condition that prevents pressure application (arterial insufficiency, pressure intolerance, etc.)
* Not having received conservative treatment for lymphedema for at least 6 months

Exclusion Criteria:

* Having history of metastases
* Having radiogenic fibrosis in the abdomino-pelvic region
* Having additional orthopedic (scoliosis, etc.), neurological (multiple sclerosis, stroke, etc.) and rheumatological diseases (ankylosing spondylitis, rheumatoid arthritis, etc.) that will affect lower extremity functions
* Having connective tissue disease that will affect tissue properties
* Having diseases (cardiac edema, peripheral artery disease, etc.) that prevent MLD and/or bandage application
* Continuation of Radiotherapy (Must have ended at least 3 months ago) and Chemotherapy applications
* Using sedatives and/or muscle relaxants that may alter muscle tone.
* Having any surgical intervention for lymphedema
* Being diagnosed with obesity (BMI>30)

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Data Record | Baseline
  Demographic, clinical and lymphedema-related data will be recorded with face-to-face interviews.
Leg circumference measurement | Change from baseline leg circumference measurement at week 3 and week 7.
  Both leg circumference measurements will be taken at 4 cm intervals from the medial malleolus. These values will then be converted to volumetric measurement using the ACOLS Limb Volume Calculation program.
Functional Evaluation | Change from baseline Lower Extremity Functional Scale at week 3 and week 7.
  The Lower Extremity Functional Scale will be used to determine the functional levels of individuals. The lower extremity functional scale consists of 20 items. Each item is scored between 0-4 and evaluated in 5 options. These options are: extreme difficulty/inability to perform the activity, quite difficult, moderate difficulty, a little difficulty and no difficulty. The total score ranges from 0-80, with higher scores representing better functional level. Individuals will be asked to mark the difficulties they have experienced or will experience in activities related to the cause of lymphedema, and the total score will be calculated.
Evaluation of Sleep Quality | Change from baseline Pittsburgh Sleep Quality Index at week 3 and week 7.
  It will be assessed by the Pittsburgh Sleep Quality Index, which evaluates the sleep quality of the individual for the last month, includes a total of 24 questions. 19 of these are self-report questions and are answered by the patient himself. Five questions are answered by the patient's spouse or roommate and are used for clinical information only and are not included in the scoring. Each question is evaluated with a number from 0 to 3. The sum of the scores of the seven components gives the total score. Sleep quality of those with a total score of 5 or less was "good"; Those with a score above 5 are considered to have "poor" sleep quality.
Evaluation of Quality of Life | Change from baseline Lymphedema Quality of Life Questionnaire at week 3 and week 7.
  The disease-specific quality of life of individuals will be evaluated using the Lymphedema Quality of Life Questionnaire. It is designed as two separate forms as lower extremity and upper extremity. A leg questionnaire will be applied to individuals. The questionnaire has 4 sub-dimensions: symptoms, body image, appearance, function, and mode. It contains 26 items in total. Individuals will be asked to tick the box that best describes how they feel about each of the questions, and the total score will be calculated.
Passive Tone | Change from baseline passive tone of myofascial tissues at week 3 and week 7.
  Passive Tone will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Stiffness | Change from baseline Stiffness of myofascial tissues at week 3 and week 7.
  Stiffness will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Decrement | Change from baseline Decrement of myofascial tissues at week 3 and week 7.
  Decrement will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Creep | Change from baseline Creep of myofascial tissues at week 3 and week 7.
  Creep will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.
Relaxation time | Change from baseline Relaxation time of myofascial tissues at week 3 and week 7.
  Relaxation time will be evaluated with MyotonPro digital palpation device which is a valid and reliable. In the measurements, the Myoton probe will be placed perpendicular to the fibers of the tissue to be measured and when the probe reaches a sufficient depth, 3 repetitive mechanical stimulus (15ms, 0.40N) will be given to the tissue that has pre-compressed (0.18N). Measurements were taken 3 times from each point and the average values will be used in statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Kablan, Asst. Prof., Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoshihara M, Shimono R, Tsuru S, Kitamura K, Sakuda H, Oguchi H, Hirota A. Risk factors for late-onset lower limb lymphedema after gynecological cancer treatment: A multi-institutional retrospective study. Eur J Surg Oncol. 2020 Jul;46(7):1334-1338. doi: 10.1016/j.ejso.2020.01.033. Epub 2020 Jan 31. PMID 32146054
- [Background] Borman P, Yaman A, Denizli M, Karahan S. The Reliability and Validity of Lymphedema Quality of Life Questionnaire-Leg in Turkish Patients with Lower Limb Lymphedema. Lymphat Res Biol. 2020 Feb;18(1):42-48. doi: 10.1089/lrb.2018.0048. Epub 2019 May 24. PMID 31135275
- [Background] Hruby RJ, Martinez ES. The Lymphatic System: An Osteopathic Review. Cureus. 2021 Jul 17;13(7):e16448. doi: 10.7759/cureus.16448. eCollection 2021 Jul. PMID 34422479